CLINICAL TRIAL: NCT03467165
Title: Magnetic Resonance Guided Focused Ultrasound Surgery: a Pilot Study in the Treatment of Pain Caused by Osteoarthritis - Hand and Hip, Challenging Joints
Brief Title: MRgFUS in the Treatment of Hand and Hip Osteoarthritic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: handhip@IORFus
Record Dates: First submitted 2018-02-23; First posted 2018-03-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis; Hip Osteoarthritis; Hand Osteoarthritis
Keywords: MRgFUS; Pain; Hip; Trapeziometacarpal joint; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Pain

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand ExAblate (Experimental): MRgFUS treatment of pain caused by trapeziometacarpal OA (and/or scaphotrapezial OA)
  Interventions: Device: MRgFUS treatment
- Hip ExAblate (Experimental): MRgFUS treatment of pain caused by hip OA
  Interventions: Device: MRgFUS treatment

INTERVENTIONS:
Device: MRgFUS treatment — MRgFUS treatment of pain caused by trapeziometacarpal OA (and/or scaphotrapezial OA)
  Arms: Hand ExAblate
Device: MRgFUS treatment — MRgFUS treatment of pain caused by hip OA
  Arms: Hip ExAblate

SUMMARY:
This project aims at performing a pilot study to provide data on safety and potential efficacy of Magnetic Resonance guided Focused Ultrasound Surgery (MRgFUS) in the treatment of pain caused by trapeziometacarpal osteoarthritis (OA) and/or scaphotrapezial OA, and by hip OA, while exploring the potential application of MRgFUS to two different and central joints burdened by OA.

DETAILED DESCRIPTION:
Pain caused by osteoarthritis is a matter of huge impact, in terms of quality of life, social and economic burden. Global aging of the population is going to worsen the problem. The hand is the most affected site in the upper limb, and involvement of the trapeziometacarpal joint is highly prevalent, with significant limitation of functionality when it happens. In the lower limb, the hip and the knee share the leading position in the clinical scenario, with the former being historically the most frequently submitted to joint replacement.

At any site, the vast majority of joint replacement surgery procedures are performed because of pain. MRgFUS has recently demonstrated a great potential in treating pain caused by different medical conditions, including osteoarthritis. The aim of the work is to study the feasibility, the safety and the potential efficacy of MRgFUS in treating pain from osteoarthritis in two "hot" spots: the hip and the trapeziometacarpal/scaphotrapezial joint.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged between 45 and 90 years
* Presence of activity-related joint pain
* Patients who have either no morning joint-related stiffness or morning stiffness that lasts no longer than 30 minutes
* Patients who have not responded to previous treatments,
* Patients with a baseline pain intensity of 4 to 8 on a 10-cm VAS
* Patients who are not candidates for immediate surgery
* Signed statement of informed consent (approved by Ethics Committee)

Exclusion Criteria:

* Prior surgery or previous local treatment (infiltration, other) in the past 3 months
* Changes in medications used during the previous 2 months
* Intravenous drug use
* Corticosteroid use of more than 3 months within the preceding year
* Diagnosis of other rheumatologic disorders
* Trauma, fracture, or osteomyelitis of the investigated joints within the preceding year
* Any neurological disease or disorders potentially affecting pain perception
* Fibromyalgia
* Pregnancy
* Patients with large scar at skin or deeper soft tissue potentially included in the planned path of the ultrasound beam
* General contraindications to MRI and/or to anaesthesiological procedures planned for the patient
* Presence of internal hardware or devices potentially affecting MR thermometry

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-27 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Intensity from Baseline | Baseline (Day1), Week 1, 2, 3, Month 1, 2, 3, 6, 9, 12
  Changes in pain intensity from baseline will be determined by a straight horizontal 10-cm linear Visual Analog Pain Scale (VAS, scale 0-10 where 0 means 'no pain at all' and 10 means 'pain as bad as it could be').
Incidence of Treatment-Related Adverse Events (Safety and Tolerability) | Through study completion, an average of 1 year
  Collecting the number of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bazzocchi, MD, PhD, Principal Investigator — The Rizzoli Ortopaedic Institute
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided